CLINICAL TRIAL: NCT00617786
Title: Current Perception Threshold Testing for Sacral Neuuromodulation Outcomes
Brief Title: CPT Testing for Sacral Neuromodulation Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Corewell Health East (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2007-176
Record Dates: First submitted 2008-02-05; First posted 2008-02-18 (Estimated); Last update posted 2011-11-23 (Estimated); Status verified 2011-11

CONDITIONS: Incontinence
Keywords: urinary urgency; urinary frequency; urge incontinence; sacral neuromodulation therapy; urgency; frequency
MeSH Terms: conditions — Urinary Incontinence, Urge | interventions — 2-cyclohexylidenhydrazo-4-phenyl-thiazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Current Perception Threshold (CPT) Testing — During the CPT testing a catheter will be placed in the bladder. The catheter has sensors to record the body's sensation of pressure. The sensation felt will be similar to a light touch and is painless. A gel pad will be placed in the general area of the vagina to record the feeling of a light touch.

SUMMARY:
This is a prospective study. Subjects will be recruited from the urology practices of Dr. Ken Peters and Dr. Ananias Diokno at William Beaumont Hospital. Subjects will be referred to the study by the clinician recommending Sacral NeuroModulation therapy (SNM).

This pilot study is to explore the effect of SNM on sensory pathways by measuring CPT values pre and post SNM treatment.

DETAILED DESCRIPTION:
Patients will be scheduled 1-2 weeks prior to planned implantation of the SNM wire electrode (Stage 1). Patients that do not have a 50% improvement in their symptoms in Stage 1 will not go on to Stage II procedures and will not undergo further CPT testing.

After enrollment, the subjects will complete a short medical history questionnaire confirming that they meet inclusion criteria and do not fall under exclusion criteria. This will include review of recent urinalysis and/or urine culture confirming the absence of a recent urinary tract infection. Participants will be given information on the relevant CPT testing including the need for bladder/urethra catheterization as part of that testing pre and post SNM therapy.

At the baseline testing visit, subjects will undergo CPT testing using transcutaneous stimulation in the distribution of the pudendal nerve on the perineum. Subjects will undergo bladder/urethral catheterization in using standard sterile technique. Once the bladder/urethral catheter is in place CPT testing will be conducted at various frequencies of to identify the current perception thresholds of each nerve fiber.

At the conclusion of the testing the catheter will be removed and the subjects will be given a single dose of an oral antibiotic to minimize infection. This meeting and testing will require approximately 60 minutes.

Patients will undergo Stage I of the SNM procedure with their own physician at a subsequent appointment.

If subjects have a 50% improvement in their symptoms after 2 weeks with Stage 1 SNM, they will under go Stage II of the SNM procedure.

The subjects will have an appointment scheduled for their follow-up CPT testing at the clinical research office 4 to 6 weeks after the Stage II procedure. The subject will be given a urinalysis and urine culture lab slip, and will be instructed to drop a urine sample off at the lab 3 days before their scheduled appointment for testing. If their urine culture is positive, they will be given a prescription for an antibiotic and excluded from this testing. They may however be tested once their urine culture is negative, as long as it is within 2 weeks of their original post-stage 2 CPT test appointment

Subjects will undergo repeat CPT testing using transcutaneous stimulation in the distribution of the pudendal nerve on the perineum. Subjects will then undergo bladder/urethral catheterization using standard sterile technique. Once the bladder/urethral catheter is in place CPT testing will then be conducted at various frequencies to identify the current perception thresholds of each nerve fiber.

At the conclusion of the testing the catheter will be removed and the patients will be given a single dose of an oral antibiotic to minimize infection. This evaluation will require approximately 60 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Established diagnosed overactive bladder
* Scheduled to receive SMN therapy by Dr. Peters or Dr. Diokno
* Women at least 18 years of age
* Capable of giving informed consent
* Capable and willing to follow all study related procedures (e.g. bladder and urethral catheterization, answering questions during CPT testing, complete questionnaires regarding pertinent medical history).

Exclusion Criteria:

* Current Urinary tract infection
* Currently participating or have participated within the past 30 days in any clinical investigation involving or impacting urinary or renal function.
* Pregnancy or intending to become pregnant during the study
* Cannot independently comprehend and complete relevant medical history questionnaires.
* The subject is deemed unsuitable for enrollment in this study by the investigators based on their history.
* Men are excluded
* TENS, PTNS or acupuncture therapy currently being used for symptoms

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2008-10; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the change in CPT measurement after placement of SNM therapy as compared to baseline CPT measurements. | visit 1

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Peters, M.D., Principal Investigator — Corewell Health East
Locations (1):
- William Beaumont Hospital, Royal Oak, Michigan, United States